CLINICAL TRIAL: NCT00568321
Title: A PHASE II RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER, PARALLEL GROUP, PROOF OF CONCEPT STUDY OF THE ANALGESIC EFFECTS OF RN624 IN ADULT PATIENTS WITH POST-HERPETIC NEURALGIA
Brief Title: RN624 For Pain Of Post-Herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A4091005; PHN POC (Other: Alias Study Number)
Record Dates: First submitted 2007-12-03; First posted 2007-12-06 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-02

CONDITIONS: Neuralgia, Postherpetic
Keywords: monoclonal antibody
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: RN624
- 2 (Active Comparator)
  Interventions: Drug: RN624
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RN624 — 50 mcg/kg
  Arms: 1
Drug: RN624 — 200 mcg/kg
  Arms: 2
Drug: Placebo — placebo
  Arms: 3

SUMMARY:
This study will test the efficacy and safety of two doses levels of RN624 versus placebo for the relief of pain caused by post-herpetic neuralgia (PHN).

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race, at least 18 years of age.
* Patients must have pain present for more than 3 months after healing of the herpes zoster skin rash.
* Has a pain score at screening that qualifies.
* Completes at least 3 average daily pain diaries during the 3 days prior to randomization and has an average pain level that qualifies.
* Body Mass Index less than or equal to 39 kg/m2.
* If female, is post-menopausal, surgically sterile, or uses adequate contraception consisting of 2 forms of birth control, one of which must be barrier method, is not lactating, and is not breastfeeding.
* Male patients must agree that female spouses/partners will use contraception as defined above or be of nonchildbearing potential (post-menopausal or surgically sterile).
* Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Patients must consent in writing to participate in the study.

Exclusion Criteria:

* Patients who cannot discontinue the use of other pain medications during the screening period and during the study.
* Disqualifying scores on questionnaires.
* Other moderate to severe pain from other conditions.
* History of allergic or anaphylactic reaction to antibodies.
* Use of biologics, including any live vaccines within 3 months of the week prior to the baseline visit.
* Unable to use acetaminophen.
* Disqualify laboratory values, Hepatitis B or C or HIV.
* Patients that have had a stroke or TIAs, dementia, epilepsy or seizures, or peripheral neuropathy from other conditions.
* Significant cardiac disease within 3 months of the study such as angina, heart attack, congestive heart failure, and other cardiac problems.
* Cancer other than basal cell or squamous cell carcinoma.
* Fails a urine test for illegal drugs including prescription drugs without a prescription.
* Plans for surgery during the study.
* History of alcoholism or drug abuse in the past two years.
* Surgery for post-herpetic neuralgia.
* Any condition that the investigator feels would put the safety of the patient at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2007-12-19 (Actual); Primary Completion 2008-12-20 (Actual); Study Completion 2009-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (31):
  - Anniston Medical Clinic/Pinnacle Research Group LLC, Anniston, Alabama
  - Anniston Neurology & Headache Mgmt. Ctr., Anniston, Alabama
  - Dedicated Clinical Research, Inc., Litchfield Park, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Jem Research, LLC, Atlantis, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Innovative Research of West Florida, Inc., Largo, Florida
  - Miami Medical Associates, Miami, Florida
  - Palm Beach Neurological Center, Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - Meridien Research, Tampa, Florida
  - Cotton-O'Neil Clinical Research, Topeka, Kansas
  - Cotton-O'Neil Clinic, Topeka, Kansas
  - International Research Center, Towson, Maryland
  - Infinity Medical Research, Inc., North Dartmouth, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Medical Advanced Pain Specialists (MAPS), Edina, Minnesota
  - A & A Pain Institute, St Louis, Missouri
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Allegheny Pain Management, PC, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - DiscoveResearch Incorporated, Bryan, Texas
  - Neurological Clinic of Texas, Dallas, Texas
  - Mobley Research Center, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Jay Ellis Jr., MD-Tejas Anesthesia, San Antonio, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - National Clinical Research, Incorporated, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Bramson C, Herrmann DN, Carey W, Keller D, Brown MT, West CR, Verburg KM, Dyck PJ. Exploring the role of tanezumab as a novel treatment for the relief of neuropathic pain. Pain Med. 2015 Jun;16(6):1163-76. doi: 10.1111/pme.12677. Epub 2015 Jan 16. PMID 25594611
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091005&StudyName=RN624%20For%20Pain%20Of%20Post-Herpetic%20Neuralgia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received single intravenous (IV) infusion of placebo matched to tanezumab (RN624 or PF-04383119) at Baseline (Day 1).
- Tanezumab 50 mcg/kg: Participants received single IV infusion of Tanezumab (RN624 or PF 04383119) 50 microgram per kilogram (mcg/kg) at Baseline (Day 1).
- Tanezumab 200 mcg/kg: Participants received single IV infusion of Tanezumab (RN624 or PF 04383119) 200 mcg/kg at Baseline (Day 1).
Period: Overall Study
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Started | 33 | 33 | 33
Treated | 31 | 33 | 32
Completed | 20 | 28 | 24
Not Completed | 13 | 5 | 9
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 8 | 5 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Randomized, not treated | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received the day 1 IV infusion (either tanezumab or placebo infusion).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg | Total
Number analyzed (Participants) | 31 | 33 | 32 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (8.7) | 71.9 (8.5) | 65.9 (14.6) | 69.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 15 | 44
  Male | 18 | 17 | 17 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Pain Numeric Rating Scale (NRS) Score at Week 6
Description: Participants assessed their average daily pain during the past 24 hours on an 11--point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain. Week 6 score was calculated as the mean of average daily pain NRS scores over the past 7 days. The change from baseline was calculated using difference between Week 6 mean score and Baseline mean score.
Time Frame: Baseline, Week 6
Population: Intent-to-treat (ITT) population included all randomized participants who received the Day 1 IV infusion (either tanezumab or placebo). Here, "number analyzed (n)" signifies those participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Baseline | 6.40 (1.55) | 6.42 (1.57) | 6.39 (1.58)
  Change at Week 6: number analyzed (Participants) | 25 | 29 | 27
  Change at Week 6 | -1.22 (1.72) | -0.97 (1.20) | -1.72 (2.40)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 50 mcg/kg; Least square (LS) mean difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.687, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean difference = 0.21, 90% CI 2-sided [-0.50 to 0.92], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 200 mcg/kg; LS mean difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.111, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean difference = -0.53, 90% CI 2-sided [-1.25 to 0.19], Standard Error of Mean 0.44

2. Secondary Outcome: Change From Baseline in Average Daily Pain Numeric Rating Scale (NRS) Score at Weeks 1, 2, 4, 8, 12 and 16
Description: Participants assessed their average daily pain during the past 24 hours on an 11--point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain. Post Baseline weekly scores were calculated as the mean of average daily pain NRS scores over the past 7 days prior to corresponding week visits. The change from baseline was calculated using difference between post baseline weekly mean score and the Baseline mean score.
Time Frame: Baseline, Week 1, 2, 4, 8, 12, 16
Population: ITT population included all randomized participants who received the Day 1 IV infusion (either tanezumab or placebo). Here, "number analyzed" signifies those participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Change at Week 1 | -0.54 (1.25) | -0.64 (1.19) | -0.91 (1.36)
  Change at Week 2: number analyzed (Participants) | 31 | 31 | 30
  Change at Week 2 | -0.80 (1.65) | -0.46 (1.42) | -0.66 (1.73)
  Change at Week 4: number analyzed (Participants) | 27 | 30 | 30
  Change at Week 4 | -1.30 (1.61) | -0.97 (1.15) | -1.46 (1.91)
  Change at Week 8: number analyzed (Participants) | 23 | 28 | 26
  Change at Week 8 | -1.18 (1.47) | -1.10 (1.36) | -1.72 (2.34)
  Change at Week 12: number analyzed (Participants) | 23 | 27 | 25
  Change at Week 12 | -1.13 (1.46) | -1.49 (1.66) | -1.45 (2.44)
  Change at Week 16: number analyzed (Participants) | 18 | 23 | 21
  Change at Week 16 | -1.18 (1.61) | -1.70 (1.78) | -1.76 (2.47)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 1: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.399, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.11, 90% CI 2-sided [-0.79 to 0.58], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.189, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.37, 90% CI 2-sided [-1.06 to 0.32], Standard Error of Mean 0.42
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 2: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.802, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.35, 90% CI 2-sided [-0.33 to 1.04], Standard Error of Mean 0.42
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.582, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.09, 90% CI 2-sided [-0.61 to 0.78], Standard Error of Mean 0.42
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 4: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.789, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.34, 90% CI 2-sided [-0.36 to 1.04], Standard Error of Mean 0.42
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.290, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.24, 90% CI 2-sided [-0.94 to 0.47], Standard Error of Mean 0.42
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 8: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.568, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.08, 90% CI 2-sided [-0.65 to 0.81], Standard Error of Mean 0.44
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.116, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.54, 90% CI 2-sided [-1.27 to 0.20], Standard Error of Mean 0.45
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 12: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.218, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.36, 90% CI 2-sided [-1.11 to 0.40], Standard Error of Mean 0.46
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority; p = 0.261, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.30, 90% CI 2-sided [-1.06 to 0.47], Standard Error of Mean 0.46
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 16: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.252, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.32, 90% CI 2-sided [-1.11 to 0.47], Standard Error of Mean 0.48
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority; p = 0.182, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.45, 90% CI 2-sided [-1.26 to 0.36], Standard Error of Mean 0.49

3. Secondary Outcome: Change From Baseline in Average Daily Pain Numeric Rating Scale (NRS) Score Over Weeks 1 to 4, 1 to 8, 1 to 12, 1 to 16, 5 to 8, 5 to 12 and 5 to 16
Description: Participants assessed their average daily pain during the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain. Scores for each time interval over the weeks were calculated from the mean of daily pain score of participants over that specified duration. Change from baseline was calculated as the average of each specified week interval (Week 1 to 4, 1 to 8, 1 to 12, 5 to 8, 5 to 12 and 5 to 16) values minus the baseline value.
Time Frame: Baseline, Week 1 to 4, Week 1 to 8, Week 1 to 12, Week 1 to 16, Week 5 to 8, Week 5 to 12, Week 5 to 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Weeks 1 to 4 | -0.87 (1.43) | -0.70 (1.13) | -1.08 (1.53)
  Weeks 1 to 8 | -0.97 (1.37) | -0.81 (1.03) | -1.35 (1.74)
  Weeks 1 to 12 | -1.01 (1.25) | -0.97 (1.07) | -1.38 (1.75)
  Weeks 1 to 16 | -1.02 (1.17) | -1.03 (1.16) | -1.43 (1.81)
  Weeks 5 to 8: number analyzed (Participants) | 25 | 29 | 29
  Weeks 5 to 8 | -1.18 (1.50) | -1.01 (1.15) | -1.61 (2.21)
  Weeks 5 to 12: number analyzed (Participants) | 25 | 29 | 29
  Weeks 5 to 12 | -1.19 (1.34) | -1.20 (1.27) | -1.50 (2.08)
  Weeks 5 to 16: number analyzed (Participants) | 25 | 29 | 29
  Weeks 5 to 16 | -1.19 (1.27) | -1.25 (1.38) | -1.52 (2.13)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 50 mcg/kg; Weeks 1 to 4: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.683, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.19, 90% CI 2-sided [-0.46 to 0.84], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.310, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.20, 90% CI 2-sided [-0.85 to 0.46], Standard Error of Mean 0.40
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 50 mcg/kg; Weeks 1 to 8: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.668, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.16, 90% CI 2-sided [-0.46 to 0.78], Standard Error of Mean 0.37
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.165, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.37, 90% CI 2-sided [-0.99 to 0.26], Standard Error of Mean 0.38
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 50 mcg/kg; Weeks 1 to 12: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.546, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.04, 90% CI 2-sided [-0.55 to 0.64], Standard Error of Mean 0.36
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.190, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.32, 90% CI 2-sided [-0.92 to 0.28], Standard Error of Mean 0.36
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 50 mcg/kg; Weeks 1 to 16: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.467, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.03, 90% CI 2-sided [-0.60 to 0.55], Standard Error of Mean 0.35
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.153, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.36, 90% CI 2-sided [-0.94 to 0.22], Standard Error of Mean 0.35
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 50 mcg/kg; Weeks 5 to 8: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.632, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.14, 90% CI 2-sided [-0.54 to 0.81], Standard Error of Mean 0.41
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; p = 0.094, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.54, 90% CI 2-sided [-1.22 to 0.14], Standard Error of Mean 0.41
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 50 mcg/kg; Weeks 5 to 12: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.468, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.03, 90% CI 2-sided [-0.68 to 0.61], Standard Error of Mean 0.39
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 3, analysis 11]; Test type: Superiority; p = 0.167, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.38, 90% CI 2-sided [-1.03 to 0.27], Standard Error of Mean 0.39
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 50 mcg/kg; Weeks 5 to 16: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.394, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.10, 90% CI 2-sided [-0.72 to 0.52], Standard Error of Mean 0.37
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p = 0.138, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.41, 90% CI 2-sided [-1.04 to 0.21], Standard Error of Mean 0.38

4. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory-Short Form (mBPI-sf) Scale Score for Worst Pain, Average Pain and Pain Severity at Weeks 1, 2, 4, 6, 8 ,12 and 16
Description: mBPI-sf is a self-administered questionnaire (5 questions) to assess pain severity and impact of pain on daily functions. Questions 1 to 4 measure the magnitude of pain (Q1 for worst, Q2 for least, Q3 for average and Q4 for pain right now) on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicate less pain. Question 5 consists of 7 item subsets which measure the level of interference of pain on daily functions: 1: general activity, 2: mood, 3: walking ability, 4: normal work, 5: relations with other, 6: sleep, 7: enjoyment of life. Each item assessed on an 11-point NRS ranging from 0 (no interference) to 10 (complete interference), where lower scores indicate less interference of pain. Pain severity score was derived from the sum of responses of questions 1-4 and ranged from 0 (no pain) to 40 (worst possible pain) with lower scores indicates less pain. Results are reported for worst pain score, average pain score and pain severity score.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8 ,12, 16
Population: ITT population included all randomized participants who received Day 1 IV infusion (either tanezumab or placebo). Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 30 | 32 | 30
units on a scale
  Baseline: Worst Pain | 7.13 (1.57) | 6.78 (1.79) | 6.93 (1.48)
  Baseline: Average Pain | 6.27 (1.46) | 6.06 (1.72) | 6.20 (1.58)
  Baseline: Pain Severity | 24.77 (6.43) | 23.78 (7.23) | 23.87 (5.90)
  Change at Week 1: Worst Pain: number analyzed (Participants) | 29 | 28 | 28
  Change at Week 1: Worst Pain | -1.10 (2.08) | -0.57 (2.22) | -0.71 (1.58)
  Change at Week 1: Average Pain: number analyzed (Participants) | 29 | 28 | 28
  Change at Week 1: Average Pain | -0.83 (1.54) | -0.46 (1.43) | -0.79 (1.55)
  Change at Week 1: Pain Severity: number analyzed (Participants) | 29 | 28 | 28
  Change at Week 1: Pain Severity | -3.59 (7.06) | -1.82 (6.42) | -2.79 (6.64)
  Change at Week 2: Worst Pain: number analyzed (Participants) | 26 | 29 | 26
  Change at Week 2: Worst Pain | -1.38 (2.14) | -0.52 (1.92) | -0.96 (2.51)
  Change at Week 2: Average Pain: number analyzed (Participants) | 26 | 29 | 26
  Change at Week 2: Average Pain | -1.19 (1.72) | -0.41 (1.18) | -0.85 (2.24)
  Change at Week 2: Pain Severity: number analyzed (Participants) | 26 | 29 | 26
  Change at Week 2: Pain Severity | -5.31 (7.17) | -1.86 (5.88) | -3.58 (9.38)
  Change at Week 4: Worst Pain: number analyzed (Participants) | 25 | 28 | 28
  Change at Week 4: Worst Pain | -1.44 (2.26) | -0.93 (1.15) | -1.18 (2.21)
  Change at Week 4: Average Pain: number analyzed (Participants) | 25 | 28 | 28
  Change at Week 4: Average Pain | -1.44 (1.64) | -0.75 (1.04) | -1.39 (2.11)
  Change at Week 4: Pain Severity: number analyzed (Participants) | 25 | 28 | 28
  Change at Week 4: Pain Severity | -5.68 (7.40) | -3.82 (4.26) | -5.21 (8.80)
  Change at Week 6: Worst Pain: number analyzed (Participants) | 21 | 27 | 25
  Change at Week 6: Worst Pain | -1.24 (1.76) | -0.93 (1.57) | -1.76 (2.74)
  Change at Week 6: Average Pain: number analyzed (Participants) | 21 | 27 | 25
  Change at Week 6: Average Pain | -1.19 (1.63) | -0.78 (1.34) | -1.72 (2.39)
  Change at Week 6: Pain Severity: number analyzed (Participants) | 21 | 27 | 25
  Change at Week 6: Pain Severity | -4.57 (5.81) | -4.07 (4.95) | -7.00 (10.39)
  Change at Week 8: Worst Pain: number analyzed (Participants) | 20 | 27 | 26
  Change at Week 8: Worst Pain | -2.00 (1.56) | -1.26 (2.09) | -1.81 (3.16)
  Change at Week 8: Average Pain: number analyzed (Participants) | 20 | 27 | 26
  Change at Week 8: Average Pain | -1.60 (1.54) | -0.96 (1.43) | -1.77 (2.44)
  Change at Week 8: Pain Severity: number analyzed (Participants) | 20 | 27 | 26
  Change at Week 8: Pain Severity | -7.60 (5.22) | -5.04 (5.78) | -6.65 (10.55)
  Change at Week 12: Worst Pain: number analyzed (Participants) | 21 | 24 | 25
  Change at Week 12: Worst Pain | -1.67 (1.49) | -1.50 (2.09) | -1.64 (3.28)
  Change at Week 12: Average Pain: number analyzed (Participants) | 21 | 24 | 25
  Change at Week 12: Average Pain | -1.38 (1.50) | -1.17 (1.49) | -1.56 (2.45)
  Change at Week 12: Pain Severity: number analyzed (Participants) | 21 | 24 | 25
  Change at Week 12: Pain Severity | -5.76 (6.03) | -5.83 (7.24) | -5.60 (10.38)
  Change at Week 16: Worst Pain: number analyzed (Participants) | 20 | 24 | 21
  Change at Week 16: Worst Pain | -1.90 (1.37) | -1.63 (2.26) | -2.38 (3.06)
  Change at Week 16: Average Pain: number analyzed (Participants) | 20 | 24 | 21
  Change at Week 16: Average Pain | -1.50 (1.28) | -1.25 (1.78) | -1.95 (2.62)
  Change at Week 16: Pain Severity: number analyzed (Participants) | 20 | 24 | 21
  Change at Week 16: Pain Severity | -6.40 (4.91) | -6.17 (7.95) | -8.38 (10.21)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 1 (Worst pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.764, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.39, 90% CI 2-sided [-0.51 to 1.30], Standard Error of Mean 0.55
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.750, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.37, 90% CI 2-sided [-0.54 to 1.28], Standard Error of Mean 0.55
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 1 (Average pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.734, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.28, 90% CI 2-sided [-0.46 to 1.03], Standard Error of Mean 0.45
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.514, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.02, 90% CI 2-sided [-0.73 to 0.77], Standard Error of Mean 0.45
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 1 (Pain severity): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.765, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 1.37, 90% CI 2-sided [-1.76 to 4.50], Standard Error of Mean 1.89
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.646, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.71, 90% CI 2-sided [-2.43 to 3.86], Standard Error of Mean 1.90
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 2 (Worst pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.895, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.69, 90% CI 2-sided [-0.22 to 1.60], Standard Error of Mean 0.55
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority; p = 0.776, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.42, 90% CI 2-sided [-0.50 to 1.34], Standard Error of Mean 0.56
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 2 (Average pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.944, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.72, 90% CI 2-sided [-0.03 to 1.47], Standard Error of Mean 0.45
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 9]; Test type: Superiority; p = 0.835, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.45, 90% CI 2-sided [-0.31 to 1.21], Standard Error of Mean 0.46
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 2 (Pain severity): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.955, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 3.23, 90% CI 2-sided [0.09 to 6.37], Standard Error of Mean 1.90
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 11]; Test type: Superiority; p = 0.884, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 2.31, 90% CI 2-sided [-0.88 to 5.49], Standard Error of Mean 1.93
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 4 (Worst pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.737, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.36, 90% CI 2-sided [-0.57 to 1.28], Standard Error of Mean 0.56
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority; p = 0.628, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.18, 90% CI 2-sided [-0.74 to 1.11], Standard Error of Mean 0.56
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 4 (Average pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.925, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.67, 90% CI 2-sided [-0.10 to 1.43], Standard Error of Mean 0.46
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.518, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.02, 90% CI 2-sided [-0.75 to 0.79], Standard Error of Mean 0.46
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 4 (Pain severity): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.810, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 1.70, 90% CI 2-sided [-1.49 to 4.88], Standard Error of Mean 1.93
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority; p = 0.600, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.49, 90% CI 2-sided [-2.72 to 3.70], Standard Error of Mean 1.94
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 6 (Worst pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.651, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.22, 90% CI 2-sided [-0.73 to 1.18], Standard Error of Mean 0.58
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 19]; Test type: Superiority; p = 0.342, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.24, 90% CI 2-sided [-1.21 to 0.73], Standard Error of Mean 0.59
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 6 (Average pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.768, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.35, 90% CI 2-sided [-0.44 to 1.14], Standard Error of Mean 0.48
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 21]; Test type: Superiority; p = 0.211, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.39, 90% CI 2-sided [-1.19 to 0.41], Standard Error of Mean 0.48
Statistical Analysis 23: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 6 (Pain severity): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.610, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.56, 90% CI 2-sided [-2.73 to 3.85], Standard Error of Mean 1.99
Statistical Analysis 24: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 23]; Test type: Superiority; p = 0.241, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -1.43, 90% CI 2-sided [-4.76 to 1.91], Standard Error of Mean 2.02
Statistical Analysis 25: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 8 (Worst pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.789, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.48, 90% CI 2-sided [-0.50 to 1.45], Standard Error of Mean 0.59
Statistical Analysis 26: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 25]; Test type: Superiority; p = 0.570, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.11, 90% CI 2-sided [-0.88 to 1.09], Standard Error of Mean 0.60
Statistical Analysis 27: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 8 (Average pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.782, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.38, 90% CI 2-sided [-0.43 to 1.19], Standard Error of Mean 0.49
Statistical Analysis 28: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 27]; Test type: Superiority; p = 0.295, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.27, 90% CI 2-sided [-1.08 to 0.55], Standard Error of Mean 0.49
Statistical Analysis 29: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 8 (Pain severity): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.804, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 1.75, 90% CI 2-sided [-1.62 to 5.11], Standard Error of Mean 2.04
Statistical Analysis 30: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.655, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.82, 90% CI 2-sided [-2.58 to 4.22], Standard Error of Mean 2.06
Statistical Analysis 31: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 12 (Worst pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.409, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.14, 90% CI 2-sided [-1.13 to 0.86], Standard Error of Mean 0.60
Statistical Analysis 32: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 31]; Test type: Superiority; p = 0.482, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.03, 90% CI 2-sided [-1.03 to 0.97], Standard Error of Mean 0.61
Statistical Analysis 33: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 12 (Average pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.592, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.12, 90% CI 2-sided [-0.71 to 0.94], Standard Error of Mean 0.50
Statistical Analysis 34: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority; p = 0.368, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.17, 90% CI 2-sided [-1.00 to 0.66], Standard Error of Mean 0.50
Statistical Analysis 35: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 12 (Pain severity): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.396, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.55, 90% CI 2-sided [-3.98 to 2.88], Standard Error of Mean 2.08
Statistical Analysis 36: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 35]; Test type: Superiority; p = 0.545, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.24, 90% CI 2-sided [-3.21 to 3.69], Standard Error of Mean 2.09
Statistical Analysis 37: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 16 (Worst pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.486, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.02, 90% CI 2-sided [-1.04 to 1.00], Standard Error of Mean 0.62
Statistical Analysis 38: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 37]; Test type: Superiority; p = 0.324, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.29, 90% CI 2-sided [-1.33 to 0.75], Standard Error of Mean 0.63
Statistical Analysis 39: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 16 (Average pain): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.563, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.08, 90% CI 2-sided [-0.76 to 0.92], Standard Error of Mean 0.51
Statistical Analysis 40: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 39]; Test type: Superiority; p = 0.282, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.30, 90% CI 2-sided [-1.16 to 0.56], Standard Error of Mean 0.52
Statistical Analysis 41: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 16 (Pain severity): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.409, Repeated Measures Model — P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.49, 90% CI 2-sided [-3.99 to 3.01], Standard Error of Mean 2.12
Statistical Analysis 42: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 4, analysis 41]; Test type: Superiority; p = 0.293, Repeated Measures Model — P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -1.18, 90% CI 2-sided [-4.76 to 2.39], Standard Error of Mean 2.17

5. Secondary Outcome: Number of Participants With Mean Average Daily Pain Score of Less Than or Equal to (<=) 2 at Weeks 1, 2, 4, 6, 8, 12 and 16
Description: Participants assessed their average daily pain during the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain. Post-baseline weekly scores were calculated as the mean of average daily pain NRS scores over the past 7 days for each specified time point. Number of participants with average daily pain score of <=2 were reported.
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants
  Week 1 | 0 | 2 | 1
  Week 2: number analyzed (Participants) | 31 | 31 | 30
  Week 2 | 1 | 2 | 1
  Week 4: number analyzed (Participants) | 27 | 30 | 30
  Week 4 | 1 | 0 | 2
  Week 6: number analyzed (Participants) | 25 | 29 | 27
  Week 6 | 2 | 2 | 7
  Week 8: number analyzed (Participants) | 23 | 28 | 26
  Week 8 | 2 | 1 | 6
  Week 12: number analyzed (Participants) | 23 | 27 | 25
  Week 12 | 3 | 4 | 4
  Week 16: number analyzed (Participants) | 18 | 23 | 21
  Week 16 | 2 | 4 | 4

6. Secondary Outcome: Number of Participants With Percent Reduction From Baseline in Average Daily Pain Score at Week 6
Description: Participants assessed their average daily pain during the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain. Week 6 score was calculated as the mean of average daily pain NRS scores over the past 7 days for each specified time point. Number of participants with specified percentage (%) of reduction in average daily pain scores from baseline at Week 6 were reported. Participants were counted more than once in different categories.
Time Frame: Baseline, Week 6
Population: ITT population included all randomized participants who received the Day 1 IV infusion (either tanezumab or placebo). Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants
  Greater than 0% reduction | 19 | 22 | 19
  Greater than or equal to (>=)10% reduction | 15 | 15 | 17
  >=20% reduction | 13 | 11 | 14
  >=30% reduction | 7 | 7 | 12
  >=40% reduction | 5 | 4 | 11
  >=50% reduction | 4 | 3 | 8
  >=60% reduction | 3 | 2 | 6
  >=70% reduction | 1 | 0 | 5
  >=80% reduction | 1 | 0 | 2
  >=90% reduction | 0 | 0 | 1
  100% reduction | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With at Least 30 Percent (%) and 50% Sustained Reduction From Baseline in Daily Average Pain Score at Week 6
Description: Participants assessed their average daily pain during the past 24 hours on an 11--point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain. Week 6 score was calculated as the mean of average daily pain NRS scores over the past 7 days before Week 6 visit. Number of participants with >=30% or >=50% of sustained reduction (defined as reduction that was maintained for a minimum duration of 4 consecutive days) in average daily pain scores from baseline at Week 6 were reported.
Time Frame: Baseline, Week 6
Population: ITT population included all randomized participants who received the Day 1 IV infusion (either tanezumab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants
  >=30% reduction | 14 | 14 | 16
  >=50% reduction | 11 | 9 | 13

8. Secondary Outcome: Number of Participants With at Least 30 Percent (%) and 50% Reduction From Baseline in Average Daily Pain Numeric Rating Scale (NRS) Score at Week 1, 2, 4, 6, 8, 12 and 16
Description: Participants assessed their average daily pain during the past 24 hours on an 11--point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain. Post-baseline weekly scores were calculated as the mean of average daily pain NRS scores over the past 7 days for each specified time point. Number of participants with >=30% or >=50% of reduction in average daily pain scores from baseline at Week 1, 2, 4, 6, 8, 12 and 16 were reported.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population included all randomized participants who received the Day 1 IV infusion (either tanezumab or placebo). Here, "number analyzed" signifies those participants who were evaluable at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants
  Week 1: >=30% reduction | 4 | 5 | 5
  Week 2: >=30% reduction: number analyzed (Participants) | 31 | 31 | 30
  Week 2: >=30% reduction | 6 | 4 | 6
  Week 4: >=30% reduction: number analyzed (Participants) | 27 | 30 | 30
  Week 4: >=30% reduction | 10 | 8 | 12
  Week 6: >=30% reduction: number analyzed (Participants) | 25 | 29 | 27
  Week 6: >=30% reduction | 7 | 7 | 12
  Week 8: >=30% reduction: number analyzed (Participants) | 23 | 28 | 26
  Week 8: >=30% reduction | 5 | 9 | 13
  Week 12: >=30% reduction: number analyzed (Participants) | 23 | 27 | 25
  Week 12: >=30% reduction | 7 | 10 | 10
  Week 16: >=30% reduction: number analyzed (Participants) | 18 | 23 | 21
  Week 16: >=30% reduction | 6 | 10 | 9
  Week 1: >=50% reduction | 1 | 3 | 2
  Week 2: >=50% reduction: number analyzed (Participants) | 31 | 31 | 30
  Week 2: >=50% reduction | 2 | 3 | 2
  Week 4: >=50% reduction: number analyzed (Participants) | 27 | 30 | 30
  Week 4: >=50% reduction | 4 | 2 | 6
  Week 6: >=50% reduction: number analyzed (Participants) | 25 | 29 | 27
  Week 6: >=50% reduction | 4 | 3 | 8
  Week 8: >=50% reduction: number analyzed (Participants) | 23 | 28 | 26
  Week 8: >=50% reduction | 2 | 2 | 9
  Week 12: >=50% reduction: number analyzed (Participants) | 23 | 27 | 25
  Week 12: >=50% reduction | 6 | 6 | 7
  Week 16: >=50% reduction: number analyzed (Participants) | 18 | 23 | 21
  Week 16: >=50% reduction | 4 | 6 | 6

9. Secondary Outcome: Time to Achieve at Least 30% (Percent) and 50% Sustained Reduction From Baseline in Average Daily Pain Score
Description: Time to achieve >=30% or >=50% sustained reduction from baseline (defined as reduction from baseline that was maintained for a total of 4 consecutive days) in average daily pain score was summarized using the Kaplan-Meier estimates. Participants assessed their average daily pain during the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain.
Time Frame: Baseline up to Week 16
Population: ITT population included all randomized participants who received the Day 1 IV infusion (either tanezumab or placebo). Here, "number analyzed" signifies number of participants who had sustained response.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
days
  Time to >=30% Reduction | 65.00 [1.00 to 65.00] | NA [NA to NA] — Median and full range was not estimable due to less than 50% of participants with events | 57.00 [1.00 to 57.00]
  Time to >=50% Reduction | NA [NA to NA] — Median and full range was not estimable due to less than 50% of participants with events | NA [NA to NA] — Median and full range was not estimable due to less than 50% of participants with events | NA [NA to NA] — Median and full range was not estimable due to less than 50% of participants with events

10. Secondary Outcome: Total Duration of at Least 30 Percent (%) and 50% Reduction From Baseline in Average Daily Pain Numeric Rating Scale (NRS) Score in Participants
Description: Total duration of response was defined as total number of days with a reduction of >=30% or >=50% in average daily pain score from baseline to Week 16. Participants assessed their average daily pain during the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain. Total duration with at least of >=30% or >=50% percent reduction in average daily pain NRS scores from Baseline to Week 16 were reported.
Time Frame: Baseline to Week 16
Population: ITT population included all randomized participants who received the Day 1 IV infusion (either tanezumab or placebo).
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
days
  Total duration for >=30% reduction | 8.00 (34.45) [0.00 to 103.00] | 2.00 (35.44) [0.00 to 106.00] | 14.50 (38.55) [0.00 to 107.00]
  Total duration for >=50% reduction | 0.00 (25.93) [0.00 to 81.00] | 0.00 (26.91) [0.00 to 99.00] | 2.50 (33.15) [0.00 to 100.00]

11. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory- Short Form (mBPI-sf) Score for Pain Interference With CS Score, GA Subtest and NW Subtest at Weeks 1, 2, 4, 6, 8, 12 and 16
Description: mBPI-sf:questionnaire (5 questions) to assess pain severity and impact of pain on daily functions. Questions 1-4 assess magnitude of pain(Q1 for worst, Q2 for least, Q3 for average and Q4 for pain right now) on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicate less pain. Question 5 consists 7 item subsets which assess level of interference of pain on daily functions: 1: general activity (GA),2: mood, 3: walking ability, 4: normal work (NW),5: relations with other,6: sleep, 7: enjoyment of life. Each item assessed on an 11-point NRS ranging from 0 (no interference) to 10 (complete interference), where lower scores =less interference of pain. These 7 items were averaged to obtain pain interference composite score (CS), ranging from 0 (no interference) to 10 (complete interference), where lower scores =less interference of pain. Change from baseline in mBPI-sf score for pain interference with CS score, GA subtest and NW subtest were reported.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12 and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 30 | 32 | 30
units on a scale
  Baseline: CS: number analyzed (Participants) | 30 | 32 | 29
  Baseline: CS | 3.87 (2.29) | 3.90 (2.46) | 4.67 (2.05)
  Baseline: GA | 4.13 (2.75) | 4.16 (3.09) | 4.83 (2.28)
  Baseline: NW: number analyzed (Participants) | 30 | 32 | 29
  Baseline: NW | 3.53 (2.66) | 3.75 (2.93) | 5.00 (2.56)
  Change at Week 1: CS: number analyzed (Participants) | 29 | 28 | 27
  Change at Week 1: CS | -0.86 (2.56) | -0.90 (1.24) | -0.99 (2.28)
  Change at Week 1: GA: number analyzed (Participants) | 29 | 28 | 28
  Change at Week 1: GA | -0.76 (3.12) | -0.57 (2.04) | -1.14 (2.86)
  Change at Week 1: NW: number analyzed (Participants) | 29 | 28 | 27
  Change at Week 1: NW | -0.48 (2.86) | -1.07 (1.36) | -1.48 (2.56)
  Change at Week 2: CS: number analyzed (Participants) | 26 | 29 | 25
  Change at Week 2: CS | -1.47 (2.18) | -0.69 (1.65) | -1.23 (2.67)
  Change at Week 2: GA: number analyzed (Participants) | 26 | 29 | 26
  Change at Week 2: GA | -1.58 (2.84) | -0.55 (2.29) | -1.04 (3.49)
  Change at Week 2: NW: number analyzed (Participants) | 26 | 29 | 25
  Change at Week 2: NW | -1.19 (2.76) | -0.59 (2.13) | -1.40 (2.68)
  Change at Week 4: CS: number analyzed (Participants) | 25 | 28 | 27
  Change at Week 4: CS | -1.22 (1.98) | -1.26 (1.66) | -1.54 (2.46)
  Change at Week 4: GA: number analyzed (Participants) | 25 | 28 | 28
  Change at Week 4: GA | -1.28 (2.61) | -1.18 (2.45) | -1.57 (3.35)
  Change at Week 4: NW: number analyzed (Participants) | 25 | 28 | 27
  Change at Week 4: NW | -1.04 (2.09) | -1.29 (1.98) | -1.63 (2.71)
  Change at Week 6: CS: number analyzed (Participants) | 21 | 27 | 24
  Change at Week 6: CS | -1.01 (1.60) | -1.20 (1.57) | -1.65 (2.77)
  Change at Week 6: GA: number analyzed (Participants) | 21 | 27 | 25
  Change at Week 6: GA | -1.05 (2.18) | -1.04 (2.14) | -1.36 (3.68)
  Change at Week 6: NW: number analyzed (Participants) | 21 | 27 | 24
  Change at Week 6: NW | -0.62 (2.18) | -1.15 (2.03) | -1.63 (3.15)
  Change at Week 8: CS: number analyzed (Participants) | 20 | 27 | 25
  Change at Week 8: CS | -1.37 (1.75) | -1.11 (1.83) | -1.41 (2.60)
  Change at Week 8: GA: number analyzed (Participants) | 20 | 27 | 26
  Change at Week 8: GA | -1.55 (2.28) | -1.04 (2.17) | -1.23 (3.39)
  Change at Week 8: NW: number analyzed (Participants) | 20 | 27 | 25
  Change at Week 8: NW | -1.10 (2.13) | -0.96 (2.23) | -1.52 (2.76)
  Change at Week 12: CS: number analyzed (Participants) | 21 | 24 | 24
  Change at Week 12: CS | -0.89 (1.69) | -1.07 (2.04) | -1.25 (3.25)
  Change at Week 12: GA: number analyzed (Participants) | 21 | 24 | 25
  Change at Week 12: GA | -0.86 (2.54) | -0.92 (2.36) | -0.92 (4.08)
  Change at Week 12: NW: number analyzed (Participants) | 21 | 24 | 24
  Change at Week 12: NW | -0.52 (2.34) | -1.00 (2.21) | -1.25 (3.33)
  Change at Week 16: CS: number analyzed (Participants) | 20 | 24 | 20
  Change at Week 16: CS | -1.46 (1.21) | -1.23 (2.02) | -1.82 (3.00)
  Change at Week 16: GA: number analyzed (Participants) | 20 | 24 | 21
  Change at Week 16: GA | -1.40 (1.82) | -1.21 (2.21) | -2.10 (3.77)
  Change at Week 16: NW: number analyzed (Participants) | 20 | 24 | 20
  Change at Week 16: NW | -1.30 (1.78) | -1.21 (2.26) | -1.80 (3.16)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 1 (CS): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.343, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.20, 90% CI 2-sided [-1.03 to 0.62], Standard Error of Mean 0.50
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.576, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.10, 90% CI 2-sided [-0.75 to 0.94], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 1 (GA): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.460, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.06, 90% CI 2-sided [-1.10 to 0.98], Standard Error of Mean 0.63
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.435, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.10, 90% CI 2-sided [-1.15 to 0.94], Standard Error of Mean 0.63
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 1 (NW): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.104, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.70, 90% CI 2-sided [-1.62 to 0.22], Standard Error of Mean 0.56
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.204, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.48, 90% CI 2-sided [-1.42 to 0.47], Standard Error of Mean 0.57
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 2 (CS): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.931, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.75, 90% CI 2-sided [-0.08 to 1.58], Standard Error of Mean 0.50
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p = 0.941, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.81, 90% CI 2-sided [-0.04 to 1.67], Standard Error of Mean 0.52
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 2 (GA): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.936, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.96, 90% CI 2-sided [-0.08 to 2.01], Standard Error of Mean 0.63
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.965, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 1.17, 90% CI 2-sided [0.11 to 2.23], Standard Error of Mean 0.64
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 2 (NW): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.855, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.59, 90% CI 2-sided [-0.33 to 1.51], Standard Error of Mean 0.56
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.765, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.42, 90% CI 2-sided [-0.54 to 1.38], Standard Error of Mean 0.58
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 4 (CS): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.504, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.01, 90% CI 2-sided [-0.84 to 0.85], Standard Error of Mean 0.51
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 13]; Test type: Superiority; p = 0.643, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.19, 90% CI 2-sided [-0.67 to 1.06], Standard Error of Mean 0.52
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 4 (GA): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.486, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.02, 90% CI 2-sided [-1.09 to 1.04], Standard Error of Mean 0.64
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 15]; Test type: Superiority; p = 0.600, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.16, 90% CI 2-sided [-0.91 to 1.24], Standard Error of Mean 0.65
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 4 (NW): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.418, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.12, 90% CI 2-sided [-1.05 to 0.82], Standard Error of Mean 0.57
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 17]; Test type: Superiority; p = 0.515, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.02, 90% CI 2-sided [-0.95 to 0.99], Standard Error of Mean 0.59
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 6 (CS): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.456, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.06, 90% CI 2-sided [-0.93 to 0.81], Standard Error of Mean 0.53
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 19]; Test type: Superiority; p = 0.556, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.08, 90% CI 2-sided [-0.82 to 0.97], Standard Error of Mean 0.54
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 6 (GA): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.448, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.09, 90% CI 2-sided [-1.19 to 1.02], Standard Error of Mean 0.67
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 21]; Test type: Superiority; p = 0.600, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.17, 90% CI 2-sided [-0.95 to 1.30], Standard Error of Mean 0.68
Statistical Analysis 23: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 6 (NW): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.225, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.44, 90% CI 2-sided [-1.41 to 0.52], Standard Error of Mean 0.59
Statistical Analysis 24: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 23]; Test type: Superiority; p = 0.387, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.17, 90% CI 2-sided [-1.18 to 0.83], Standard Error of Mean 0.61
Statistical Analysis 25: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 8 (CS): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.657, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.22, 90% CI 2-sided [-0.67 to 1.11], Standard Error of Mean 0.54
Statistical Analysis 26: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 25]; Test type: Superiority; p = 0.808, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.48, 90% CI 2-sided [-0.43 to 1.40], Standard Error of Mean 0.55
Statistical Analysis 27: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 8 (GA): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.742, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.45, 90% CI 2-sided [-0.68 to 1.57], Standard Error of Mean 0.68
Statistical Analysis 28: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 27]; Test type: Superiority; p = 0.923, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.99, 90% CI 2-sided [-0.16 to 2.14], Standard Error of Mean 0.70
Statistical Analysis 29: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 8 (NW): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.490, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.02, 90% CI 2-sided [-1.01 to 0.98], Standard Error of Mean 0.60
Statistical Analysis 30: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 29]; Test type: Superiority; p = 0.609, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.17, 90% CI 2-sided [-0.86 to 1.20], Standard Error of Mean 0.62
Statistical Analysis 31: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 12 (CS): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.362, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.19, 90% CI 2-sided [-1.10 to 0.71], Standard Error of Mean 0.55
Statistical Analysis 32: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 31]; Test type: Superiority; p = 0.610, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.16, 90% CI 2-sided [-0.77 to 1.09], Standard Error of Mean 0.56
Statistical Analysis 33: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 12 (GA): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.376, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.22, 90% CI 2-sided [-1.37 to 0.93], Standard Error of Mean 0.70
Statistical Analysis 34: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 33]; Test type: Superiority; p = 0.733, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.44, 90% CI 2-sided [-0.73 to 1.60], Standard Error of Mean 0.71
Statistical Analysis 35: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 12 (NW): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.303, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.32, 90% CI 2-sided [-1.33 to 0.69], Standard Error of Mean 0.61
Statistical Analysis 36: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 35]; Test type: Superiority; p = 0.548, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.08, 90% CI 2-sided [-0.97 to 1.12], Standard Error of Mean 0.63
Statistical Analysis 37: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 16 (CS): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.609, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.15, 90% CI 2-sided [-0.77 to 1.08], Standard Error of Mean 0.56
Statistical Analysis 38: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 37]; Test type: Superiority; p = 0.590, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.13, 90% CI 2-sided [-0.83 to 1.10], Standard Error of Mean 0.59
Statistical Analysis 39: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 16 (GA): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.556, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.10, 90% CI 2-sided [-1.07 to 1.27], Standard Error of Mean 0.71
Statistical Analysis 40: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 39]; Test type: Superiority; p = 0.443, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.11, 90% CI 2-sided [-1.32 to 1.11], Standard Error of Mean 0.73
Statistical Analysis 41: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 16 (NW): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.527, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.04, 90% CI 2-sided [-0.99 to 1.07], Standard Error of Mean 0.62
Statistical Analysis 42: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 11, analysis 41]; Test type: Superiority; p = 0.583, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.14, 90% CI 2-sided [-0.95 to 1.22], Standard Error of Mean 0.66

12. Secondary Outcome: Number of Participants With Change From Baseline in Patient's Global Assessment of Pain Score at Weeks 1, 2, 4, 6, 8, 12 and 16
Description: Patient's global assessment of pain from post-herpetic neuralgia assessed participant's overall impression of disease activity. Participants answered: "Considering all the ways your pain from post-herpetic neuralgia, how are you doing today?". Participants responded using a 5--point Likert scale with a score of 1 being the best (very good) and a score of 5 being the worst (very poor) with lower scores indicating better condition. Number of participants who reported a change from Baseline of -4, -3, -2, -1, 0, 1, 2, 3, 4 in Patient's Global Assessment of Pain scores at each specified time-point were presented.
Time Frame: Baseline, Week 1, 2, 4, 6, 8 ,12, 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants
  Week 1: Change= --4: number analyzed (Participants) | 29 | 29 | 27
  Week 1: Change= --4 | 0 | 0 | 0
  Week 1: Change= --3: number analyzed (Participants) | 29 | 29 | 27
  Week 1: Change= --3 | 1 | 0 | 0
  Week 1: Change= --2: number analyzed (Participants) | 29 | 29 | 27
  Week 1: Change= --2 | 3 | 1 | 0
  Week 1: Change= --1: number analyzed (Participants) | 29 | 29 | 27
  Week 1: Change= --1 | 4 | 4 | 8
  Week 1: Change= 0: number analyzed (Participants) | 29 | 29 | 27
  Week 1: Change= 0 | 15 | 19 | 11
  Week 1: Change= 1: number analyzed (Participants) | 29 | 29 | 27
  Week 1: Change= 1 | 5 | 4 | 7
  Week 1: Change= 2: number analyzed (Participants) | 29 | 29 | 27
  Week 1: Change= 2 | 1 | 1 | 0
  Week 1: Change= 3: number analyzed (Participants) | 29 | 29 | 27
  Week 1: Change= 3 | 0 | 0 | 0
  Week 1: Change= 4: number analyzed (Participants) | 29 | 29 | 27
  Week 1: Change= 4 | 0 | 0 | 1
  Week 2: Change= --4: number analyzed (Participants) | 27 | 29 | 25
  Week 2: Change= --4 | 0 | 0 | 0
  Week 2: Change= --3: number analyzed (Participants) | 27 | 29 | 25
  Week 2: Change= --3 | 1 | 0 | 0
  Week 2: Change= --2: number analyzed (Participants) | 27 | 29 | 25
  Week 2: Change= --2 | 3 | 0 | 2
  Week 2: Change= --1: number analyzed (Participants) | 27 | 29 | 25
  Week 2: Change= --1 | 5 | 7 | 2
  Week 2: Change= 0: number analyzed (Participants) | 27 | 29 | 25
  Week 2: Change= 0 | 15 | 15 | 17
  Week 2: Change= 1: number analyzed (Participants) | 27 | 29 | 25
  Week 2: Change= 1 | 2 | 7 | 3
  Week 2: Change= 2: number analyzed (Participants) | 27 | 29 | 25
  Week 2: Change= 2 | 0 | 0 | 1
  Week 2: Change= 3: number analyzed (Participants) | 27 | 29 | 25
  Week 2: Change= 3 | 1 | 0 | 0
  Week 2: Change= 4: number analyzed (Participants) | 27 | 29 | 25
  Week 2: Change= 4 | 0 | 0 | 0
  Week 4: Change= --4: number analyzed (Participants) | 25 | 28 | 27
  Week 4: Change= --4 | 0 | 0 | 0
  Week 4: Change= --3: number analyzed (Participants) | 25 | 28 | 27
  Week 4: Change= --3 | 1 | 0 | 0
  Week 4: Change= --2: number analyzed (Participants) | 25 | 28 | 27
  Week 4: Change= --2 | 1 | 1 | 1
  Week 4: Change= --1: number analyzed (Participants) | 25 | 28 | 27
  Week 4: Change= --1 | 7 | 5 | 8
  Week 4: Change= 0: number analyzed (Participants) | 25 | 28 | 27
  Week 4: Change= 0 | 10 | 20 | 16
  Week 4: Change= 1: number analyzed (Participants) | 25 | 28 | 27
  Week 4: Change= 1 | 5 | 1 | 2
  Week 4: Change= 2: number analyzed (Participants) | 25 | 28 | 27
  Week 4: Change= 2 | 0 | 1 | 0
  Week 4: Change= 3: number analyzed (Participants) | 25 | 28 | 27
  Week 4: Change= 3 | 1 | 0 | 0
  Week 4: Change= 4: number analyzed (Participants) | 25 | 28 | 27
  Week 4: Change= 4 | 0 | 0 | 0
  Week 6: Change= --4: number analyzed (Participants) | 21 | 27 | 24
  Week 6: Change= --4 | 0 | 0 | 0
  Week 6: Change= --3: number analyzed (Participants) | 21 | 27 | 24
  Week 6: Change= --3 | 0 | 0 | 0
  Week 6: Change= --2: number analyzed (Participants) | 21 | 27 | 24
  Week 6: Change= --2 | 1 | 1 | 2
  Week 6: Change= --1: number analyzed (Participants) | 21 | 27 | 24
  Week 6: Change= --1 | 6 | 7 | 6
  Week 6: Change= 0: number analyzed (Participants) | 21 | 27 | 24
  Week 6: Change= 0 | 11 | 17 | 13
  Week 6: Change= 1: number analyzed (Participants) | 21 | 27 | 24
  Week 6: Change= 1 | 3 | 0 | 2
  Week 6: Change= 2: number analyzed (Participants) | 21 | 27 | 24
  Week 6: Change= 2 | 0 | 2 | 1
  Week 6: Change= 3: number analyzed (Participants) | 21 | 27 | 24
  Week 6: Change= 3 | 0 | 0 | 0
  Week 6: Change= 4: number analyzed (Participants) | 21 | 27 | 24
  Week 6: Change= 4 | 0 | 0 | 0
  Week 8: Change= --4: number analyzed (Participants) | 20 | 27 | 25
  Week 8: Change= --4 | 0 | 0 | 0
  Week 8: Change= --3: number analyzed (Participants) | 20 | 27 | 25
  Week 8: Change= --3 | 0 | 0 | 0
  Week 8: Change= --2: number analyzed (Participants) | 20 | 27 | 25
  Week 8: Change= --2 | 1 | 1 | 2
  Week 8: Change= -1: number analyzed (Participants) | 20 | 27 | 25
  Week 8: Change= -1 | 7 | 7 | 8
  Week 8: Change= 0: number analyzed (Participants) | 20 | 27 | 25
  Week 8: Change= 0 | 9 | 17 | 12
  Week 8: Change= 1: number analyzed (Participants) | 20 | 27 | 25
  Week 8: Change= 1 | 3 | 1 | 2
  Week 8: Change= 2: number analyzed (Participants) | 20 | 27 | 25
  Week 8: Change= 2 | 0 | 1 | 1
  Week 8: Change= 3: number analyzed (Participants) | 20 | 27 | 25
  Week 8: Change= 3 | 0 | 0 | 0
  Week 8: Change= 4: number analyzed (Participants) | 20 | 27 | 25
  Week 8: Change= 4 | 0 | 0 | 0
  Week 12: Change= -4: number analyzed (Participants) | 21 | 24 | 24
  Week 12: Change= -4 | 0 | 0 | 0
  Week 12: Change= -3: number analyzed (Participants) | 21 | 24 | 24
  Week 12: Change= -3 | 0 | 0 | 1
  Week 12: Change= -2: number analyzed (Participants) | 21 | 24 | 24
  Week 12: Change= -2 | 0 | 1 | 3
  Week 12: Change= -1: number analyzed (Participants) | 21 | 24 | 24
  Week 12: Change= -1 | 6 | 6 | 5
  Week 12: Change= 0: number analyzed (Participants) | 21 | 24 | 24
  Week 12: Change= 0 | 11 | 12 | 12
  Week 12: Change= 1 | 3 | 4 | 3
  Week 12: Change= 2: number analyzed (Participants) | 21 | 24 | 24
  Week 12: Change= 2 | 1 | 1 | 0
  Week 12: Change= 3: number analyzed (Participants) | 21 | 24 | 24
  Week 12: Change= 3 | 0 | 0 | 0
  Week 12: Change= 4: number analyzed (Participants) | 21 | 24 | 24
  Week 12: Change= 4 | 0 | 0 | 0
  Week 16: Change= -4: number analyzed (Participants) | 20 | 24 | 20
  Week 16: Change= -4 | 0 | 0 | 0
  Week 16: Change= -3: number analyzed (Participants) | 20 | 24 | 20
  Week 16: Change= -3 | 0 | 0 | 1
  Week 16: Change= -2: number analyzed (Participants) | 20 | 24 | 20
  Week 16: Change= -2 | 0 | 1 | 1
  Week 16: Change= -1: number analyzed (Participants) | 20 | 24 | 20
  Week 16: Change= -1 | 5 | 5 | 6
  Week 16: Change= 0: number analyzed (Participants) | 20 | 24 | 20
  Week 16: Change= 0 | 14 | 15 | 10
  Week 16: Change= 1: number analyzed (Participants) | 20 | 24 | 20
  Week 16: Change= 1 | 1 | 2 | 2
  Week 16: Change= 2: number analyzed (Participants) | 20 | 24 | 20
  Week 16: Change= 2 | 0 | 1 | 0
  Week 16: Change= 3: number analyzed (Participants) | 20 | 24 | 20
  Week 16: Change= 3 | 0 | 0 | 0
  Week 16: Change= 4: number analyzed (Participants) | 20 | 24 | 20
  Week 16: Change= 4 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Each Response Level of Patient's Global Evaluation of Study Medication
Description: Participants provided their response for patient's global evaluation of study medication by answering a question. Participants answered: "In all ways, how would you rate your overall response to the study medication today?" Participants responded using a 4-¬point likert scale where 1 = poor, 2 = fair, 3 = good and 4 = excellent. Higher score indicating better overall response to the treatment. Number of participants with each response level (poor, fair, good and excellent) were reported.
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants
  Week 1: Poor: number analyzed (Participants) | 29 | 30 | 29
  Week 1: Poor | 11 | 13 | 13
  Week 1: Fair: number analyzed (Participants) | 29 | 30 | 29
  Week 1: Fair | 5 | 5 | 8
  Week 1: Good: number analyzed (Participants) | 29 | 30 | 29
  Week 1: Good | 11 | 9 | 7
  Week 1: Excellent: number analyzed (Participants) | 29 | 30 | 29
  Week 1: Excellent | 2 | 3 | 1
  Week 2: Poor: number analyzed (Participants) | 27 | 29 | 27
  Week 2: Poor | 7 | 12 | 13
  Week 2: Fair: number analyzed (Participants) | 27 | 29 | 27
  Week 2: Fair | 6 | 4 | 9
  Week 2: Good: number analyzed (Participants) | 27 | 29 | 27
  Week 2: Good | 11 | 11 | 4
  Week 2: Excellent: number analyzed (Participants) | 27 | 29 | 27
  Week 2: Excellent | 3 | 2 | 1
  Week 4: Poor: number analyzed (Participants) | 26 | 29 | 29
  Week 4: Poor | 7 | 7 | 7
  Week 4: Fair: number analyzed (Participants) | 26 | 29 | 29
  Week 4: Fair | 9 | 11 | 14
  Week 4: Good: number analyzed (Participants) | 26 | 29 | 29
  Week 4: Good | 8 | 10 | 6
  Week 4: Excellent: number analyzed (Participants) | 26 | 29 | 29
  Week 4: Excellent | 2 | 1 | 2
  Week 6: Poor: number analyzed (Participants) | 22 | 28 | 26
  Week 6: Poor | 7 | 8 | 7
  Week 6: Fair: number analyzed (Participants) | 22 | 28 | 26
  Week 6: Fair | 8 | 9 | 7
  Week 6: Good: number analyzed (Participants) | 22 | 28 | 26
  Week 6: Good | 5 | 11 | 7
  Week 6: Excellent: number analyzed (Participants) | 22 | 28 | 26
  Week 6: Excellent | 2 | 0 | 5
  Week 8: Poor: number analyzed (Participants) | 20 | 28 | 26
  Week 8: Poor | 4 | 9 | 10
  Week 8: Fair: number analyzed (Participants) | 20 | 28 | 26
  Week 8: Fair | 4 | 9 | 5
  Week 8: Good: number analyzed (Participants) | 20 | 28 | 26
  Week 8: Good | 10 | 8 | 7
  Week 8: Excellent: number analyzed (Participants) | 20 | 28 | 26
  Week 8: Excellent | 2 | 2 | 4
  Week 12: Poor: number analyzed (Participants) | 22 | 25 | 24
  Week 12: Poor | 7 | 8 | 10
  Week 12: Fair: number analyzed (Participants) | 22 | 25 | 24
  Week 12: Fair | 6 | 8 | 5
  Week 12: Good: number analyzed (Participants) | 22 | 25 | 24
  Week 12: Good | 9 | 7 | 5
  Week 12: Excellent: number analyzed (Participants) | 22 | 25 | 24
  Week 12: Excellent | 0 | 2 | 4
  Week 16: Poor: number analyzed (Participants) | 21 | 25 | 21
  Week 16: Poor | 3 | 6 | 6
  Week 16: Fair: number analyzed (Participants) | 21 | 25 | 21
  Week 16: Fair | 7 | 8 | 6
  Week 16: Good: number analyzed (Participants) | 21 | 25 | 21
  Week 16: Good | 8 | 7 | 5
  Week 16: Excellent: number analyzed (Participants) | 21 | 25 | 21
  Week 16: Excellent | 3 | 4 | 4

14. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory-Short Form (mBPI-sf) Score for Pain Interference With Sleep at Weeks 1, 2, 4, 6, 8 ,12 and 16
Description: mBPI-sf is a self-administered questionnaire (5 questions) to assess pain severity and impact of pain on daily functions. Questions (Q) 1-4 assess magnitude of pain severity (Q1 for worst, Q2 for least, Q3 for average, Q4 for pain right now) on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicate less pain. Question 5 consists of 7 item subsets which assess the level of interference of pain on daily functions: 1: general activity, 2: mood, 3: walking ability, 4: normal work, 5: relations with other, 6: sleep, 7: enjoyment of life. Each item was assessed on an 11-point NRS ranging from 0 (no interference) to 10 (complete interference), where lower scores indicated less interference of pain. Change from Baseline in mBPI-sf score for pain interference with sleep were reported.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12, 16
Population: ITT population included all randomized participants who received Day 1 IV infusion (either tanezumab or placebo). Here, ''overall number of participants analyzed'' signifies number of participants evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 30 | 32 | 29
units on a scale
  Baseline | 4.87 (3.06) | 4.66 (2.74) | 5.48 (2.59)
  Change at Week 1: number analyzed (Participants) | 29 | 28 | 27
  Change at Week 1 | -1.03 (3.34) | -1.50 (2.20) | -1.37 (3.21)
  Change at Week 2: number analyzed (Participants) | 26 | 29 | 25
  Change at Week 2 | -1.96 (2.68) | -1.03 (2.78) | -1.72 (3.81)
  Change at Week 4: number analyzed (Participants) | 25 | 28 | 27
  Change at Week 4 | -1.60 (2.66) | -1.71 (2.19) | -2.04 (3.13)
  Change at Week 6: number analyzed (Participants) | 21 | 27 | 24
  Change at Week 6 | -1.19 (1.72) | -1.85 (2.23) | -2.46 (3.40)
  Change at Week 8: number analyzed (Participants) | 20 | 27 | 25
  Change at Week 8 | -1.80 (1.88) | -1.81 (2.69) | -2.16 (3.41)
  Change at Week 12: number analyzed (Participants) | 21 | 24 | 24
  Change at Week 12 | -1.38 (1.96) | -1.63 (2.83) | -1.83 (4.25)
  Change at Week 16: number analyzed (Participants) | 20 | 24 | 20
  Change at Week 16 | -1.90 (1.52) | -1.71 (3.22) | -2.45 (3.72)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 50 mcg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.111, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.77, 90% CI 2-sided [-1.81 to 0.27], Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.523, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.04, 90% CI 2-sided [-1.02 to 1.09], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 50 mcg/kg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.887, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.77, 90% CI 2-sided [-0.28 to 1.81], Standard Error of Mean 0.63
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.903, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.85, 90% CI 2-sided [-0.23 to 1.92], Standard Error of Mean 0.65
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 50 mcg/kg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.472, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.05, 90% CI 2-sided [-1.11 to 1.02], Standard Error of Mean 0.64
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.628, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.22, 90% CI 2-sided [-0.87 to 1.30], Standard Error of Mean 0.66
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 6: LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.243, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.47, 90% CI 2-sided [-1.58 to 0.64], Standard Error of Mean 0.67
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority; p = 0.346, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.27, 90% CI 2-sided [-1.42 to 0.87], Standard Error of Mean 0.69
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 50 mcg/kg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.467, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.06, 90% CI 2-sided [-1.19 to 1.08], Standard Error of Mean 0.69
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.670, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.31, 90% CI 2-sided [-0.85 to 1.47], Standard Error of Mean 0.70
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 50 mcg/kg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority; p = 0.286, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.40, 90% CI 2-sided [-1.55 to 0.76], Standard Error of Mean 0.70
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority; p = 0.598, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.18, 90% CI 2-sided [-1.00 to 1.35], Standard Error of Mean 0.71
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 50 mcg/kg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority; p = 0.453, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.08, 90% CI 2-sided [-1.26 to 1.09], Standard Error of Mean 0.71
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority; p = 0.472, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.05, 90% CI 2-sided [-1.28 to 1.17], Standard Error of Mean 0.74

15. Secondary Outcome: Number of Participants Who Discontinued the Study Due to Lack of Efficacy
Time Frame: Baseline up to Week 16
Population: ITT population included all randomized participants who received the Day 1 IV infusion (either tanezumab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants | 8 | 5 | 6

16. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Time to discontinuation due to lack of efficacy was defined as the time interval from the date of study drug administration up to the date of discontinuation of participant from study due to lack of efficacy.
Time Frame: Baseline up to Week 16
Population: ITT population included all randomized participants who received the Day 1 IV infusion (either tanezumab or placebo).
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
days | 71.32 (4.95) | 40.79 (1.82) | 72.13 (3.91)

17. Secondary Outcome: Number of Participants Who Used Rescue Medications
Description: In case of inadequate pain relief for post-herpetic neuralgia, acetaminophen up to 3000 mg per day up to 3 days in a week could be taken as rescue medication. Number of participants with any use of rescue medication during the specified study week were summarized.
Time Frame: Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants
  Week 1 | 18 | 22 | 12
  Week 2: number analyzed (Participants) | 31 | 33 | 31
  Week 2 | 16 | 17 | 14
  Week 3: number analyzed (Participants) | 31 | 31 | 30
  Week 3 | 15 | 17 | 17
  Week 4: number analyzed (Participants) | 27 | 31 | 30
  Week 4 | 10 | 18 | 13
  Week 5: number analyzed (Participants) | 27 | 30 | 30
  Week 5 | 11 | 16 | 10
  Week 6: number analyzed (Participants) | 25 | 29 | 29
  Week 6 | 12 | 15 | 15
  Week 7: number analyzed (Participants) | 25 | 29 | 29
  Week 7 | 10 | 13 | 13
  Week 8: number analyzed (Participants) | 24 | 28 | 28
  Week 8 | 7 | 17 | 11
  Week 9: number analyzed (Participants) | 23 | 28 | 28
  Week 9 | 6 | 15 | 12
  Week 10: number analyzed (Participants) | 23 | 28 | 27
  Week 10 | 9 | 14 | 13
  Week 11: number analyzed (Participants) | 23 | 28 | 27
  Week 11 | 9 | 15 | 11
  Week 12: number analyzed (Participants) | 23 | 28 | 26
  Week 12 | 10 | 17 | 11
  Week 13: number analyzed (Participants) | 22 | 28 | 25
  Week 13 | 8 | 15 | 9
  Week 14: number analyzed (Participants) | 21 | 28 | 25
  Week 14 | 10 | 15 | 8
  Week 15: number analyzed (Participants) | 21 | 27 | 24
  Week 15 | 8 | 12 | 12
  Week 16: number analyzed (Participants) | 18 | 27 | 23
  Week 16 | 6 | 14 | 13

18. Secondary Outcome: Duration of Rescue Medication Use
Description: In case of inadequate pain relief for post-herpetic neuralgia, acetaminophen up to 3000 mg per day up to 3 days in a week could be taken as rescue medication. Number of days participant used rescue medication, during the specified weeks were summarized.
Time Frame: Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
days
  Week 1 | 1.00 [0.00 to 6.00] | 1.00 [0.00 to 6.00] | 0.00 [0.00 to 6.00]
  Week 2: number analyzed (Participants) | 31 | 33 | 31
  Week 2 | 1.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00]
  Week 3: number analyzed (Participants) | 31 | 31 | 30
  Week 3 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 1.50 [0.00 to 7.00]
  Week 4: number analyzed (Participants) | 27 | 31 | 30
  Week 4 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00]
  Week 5: number analyzed (Participants) | 27 | 30 | 30
  Week 5 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00]
  Week 6: number analyzed (Participants) | 25 | 29 | 29
  Week 6 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00]
  Week 7: number analyzed (Participants) | 25 | 29 | 29
  Week 7 | 0.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00]
  Week 8: number analyzed (Participants) | 24 | 28 | 28
  Week 8 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00]
  Week 9: number analyzed (Participants) | 23 | 28 | 28
  Week 9 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 0.00 [0.00 to 6.00]
  Week 10: number analyzed (Participants) | 23 | 28 | 27
  Week 10 | 0.00 [0.00 to 7.00] | 0.50 [0.00 to 7.00] | 0.00 [0.00 to 6.00]
  Week 11: number analyzed (Participants) | 23 | 28 | 27
  Week 11 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00]
  Week 12: number analyzed (Participants) | 23 | 28 | 26
  Week 12 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00]
  Week 13: number analyzed (Participants) | 22 | 28 | 25
  Week 13 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00]
  Week 14: number analyzed (Participants) | 21 | 28 | 25
  Week 14 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00]
  Week 15: number analyzed (Participants) | 21 | 27 | 24
  Week 15 | 0.00 [0.00 to 7.00] | 0.00 [0.00 to 7.00] | 0.50 [0.00 to 7.00]
  Week 16: number analyzed (Participants) | 18 | 27 | 23
  Week 16 | 0.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00] | 1.00 [0.00 to 7.00]

19. Secondary Outcome: Amount of Rescue Medication Taken
Description: In case of inadequate pain relief for post-herpetic neuralgia, acetaminophen up to 3000 mg per day up to 3 days in a week could be taken as rescue medication. The total dosage of acetaminophen (in mg) used during the specified week were summarized.
Time Frame: Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
milligram
  Week 1 | 3677.4 (5348.8) | 3015.2 (4118.3) | 2125.0 (3535.5)
  Week 2: number analyzed (Participants) | 31 | 33 | 31
  Week 2 | 3419.4 (4949.9) | 3515.2 (4752.4) | 2467.7 (4106.8)
  Week 3: number analyzed (Participants) | 31 | 31 | 30
  Week 3 | 2661.3 (4772.1) | 2774.2 (4118.7) | 3100.0 (4810.9)
  Week 4: number analyzed (Participants) | 27 | 31 | 30
  Week 4 | 2851.9 (4598.9) | 2387.1 (3874.5) | 1733.3 (3109.3)
  Week 5: number analyzed (Participants) | 27 | 30 | 30
  Week 5 | 2500.0 (4759.6) | 1900.0 (3046.8) | 1883.3 (3600.0)
  Week 6: number analyzed (Participants) | 25 | 29 | 29
  Week 6 | 2960.0 (4964.3) | 1827.6 (3282.2) | 1810.3 (3100.7)
  Week 7: number analyzed (Participants) | 25 | 29 | 29
  Week 7 | 2920.0 (5217.5) | 1758.6 (3712.0) | 1689.7 (3137.9)
  Week 8: number analyzed (Participants) | 24 | 28 | 28
  Week 8 | 1770.8 (4175.4) | 2303.6 (3432.8) | 1517.9 (2447.5)
  Week 9: number analyzed (Participants) | 23 | 28 | 28
  Week 9 | 1760.9 (4504.7) | 2160.7 (3372.1) | 1517.9 (2488.8)
  Week 10: number analyzed (Participants) | 23 | 28 | 27
  Week 10 | 1847.8 (3767.2) | 2339.3 (3768.9) | 1759.3 (2693.9)
  Week 11: number analyzed (Participants) | 23 | 28 | 27
  Week 11 | 1891.3 (3394.4) | 2446.4 (3871.4) | 1666.7 (2609.2)
  Week 12: number analyzed (Participants) | 23 | 28 | 26
  Week 12 | 2326.1 (4193.1) | 2214.3 (3486.6) | 1961.5 (3168.4)
  Week 13: number analyzed (Participants) | 22 | 28 | 25
  Week 13 | 2590.9 (4371.5) | 2142.9 (3042.5) | 1400.0 (2594.1)
  Week 14: number analyzed (Participants) | 21 | 28 | 25
  Week 14 | 2285.7 (3477.0) | 1821.4 (2385.2) | 1160.0 (2330.6)
  Week 15: number analyzed (Participants) | 21 | 27 | 24
  Week 15 | 1595.2 (3084.7) | 2129.6 (3142.7) | 1854.2 (2826.4)
  Week 16: number analyzed (Participants) | 18 | 27 | 23
  Week 16 | 916.7 (1759.4) | 1870.4 (2475.2) | 2065.2 (3145.4)

20. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 112 days after last dose (up to Week 16) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to 112 days after the last dose of study drug (up to Week 16)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants
  AEs | 20 | 24 | 21
  SAEs | 1 | 2 | 1

21. Secondary Outcome: Number of Participants With Abnormal Physical Examinations Findings at Screening
Description: Physical examination included the examination of abdomen, ears, extremities, eyes, general appearance, head, heart, lungs, musculoskeletal assessment, neck, nose, skin, throat and thyroid. Abnormalities in physical examination was based on investigator's discretion.
Time Frame: Screening visit (1 day prior to Day 1 baseline visit)
Population: Safety analysis population included all participants who received the day 1 IV infusion (either tanezumab or placebo infusion). Here, "number analyzed" signifies those participants who were evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants
  Abdomen: number analyzed (Participants) | 29 | 33 | 32
  Abdomen | 0 | 3 | 1
  Ear | 0 | 1 | 2
  Extremities: number analyzed (Participants) | 29 | 33 | 29
  Extremities | 2 | 5 | 4
  Eyes | 1 | 4 | 0
  General: number analyzed (Participants) | 31 | 33 | 31
  General | 0 | 0 | 0
  Head | 2 | 0 | 3
  Heart: number analyzed (Participants) | 29 | 33 | 32
  Heart | 1 | 3 | 1
  Lungs | 0 | 0 | 2
  Musculoskeletal: number analyzed (Participants) | 28 | 33 | 32
  Musculoskeletal | 1 | 3 | 4
  Neck | 0 | 2 | 1
  Nose | 1 | 1 | 0
  Skin: number analyzed (Participants) | 28 | 33 | 32
  Skin | 10 | 10 | 10
  Throat | 0 | 0 | 0
  Thyroid | 0 | 1 | 1

22. Secondary Outcome: Number of Participants With Change From Baseline in Physical Examinations Findings at Week 16
Description: Physical examination included the examination of abdomen, ears, extremities, eyes, general appearance, head, heart, lungs, musculoskeletal assessment, neck, nose, skin, throat and thyroid.
Time Frame: Baseline, Week 16
Population: Safety analysis population included all participants who received the day 1 IV infusion (either tanezumab or placebo infusion). Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 30 | 32 | 31
Participants | 1 | 3 | 1

23. Secondary Outcome: Number of Participants With Change From Baseline in Neurological Examination Findings at Week 16
Description: Neurological examination included the assessment of cranial nerve function, coordination, reflexes, proprioception, mental status, motor function, gait and station and sensory function (sharp sensation, warm/cold sensation, light touch, deep pressure, and vibration sensation).
Time Frame: Baseline, Week 16
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 32 | 32
Participants | 1 | 0 | 0

24. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs at Week 16
Description: Vital signs included the assessment of the following: body temperature, blood pressure, heart rate and respiratory rate. Criteria for clinically significant vital signs included: heart rate value of less than (<) 40 beats per minute and greater than (>) 150 beats per minute, systolic blood pressure (SBP) of <80 or >210 millimeter of mercury (mmHg), diastolic blood pressure (DBP) of <40 or >130 mmHg, body temperature <32 or >40 degree centigrade, respiratory rate of <10 or >50 breaths/minute.
Time Frame: Baseline, Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
Participants | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Abnormality criteria: hematology (hemoglobin; hematocrit; red blood cell count [less than {<}0.8* lower limit of normal [LLN], platelets <0.5* LLN,>1.75* upper limit of normal (ULN), white blood cell count<0.6* LLN, >1.5* ULN, liver function (total bilirubin>1.5* ULN, aspartate aminotransferase; alanine aminotransferase; gamma GT, LDH, alkaline phosphatase>3.0* ULN, total protein; albumin<0.8* LLN; >1.2* ULN), renal function (blood urea nitrogen; creatinine>1.3* ULN, uric acid>1.2* ULN), lipids (cholesterol, triglycerides >1.3*ULN), electrolytes (sodium <0.95* LLN, >1.05* ULN; potassium; chloride; calcium; magnesium; phosphate; bicarbonate<0.9* LLN, >1.1* ULN), chemistry (glucose <0.6*LLN, >1.5*ULN; creatine kinase >2.0*ULN), urinalysis (specific gravity <1.003, >1.030; pH<4.5, >8, glucose; protein; blood; ketones; urobilinogen; bilirubin; nitrite, esterase>=1).
Time Frame: Baseline up to Week 16
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 32 | 32
Participants | 22 | 25 | 20

26. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for abnormality in ECG parameters: Maximum corrected QT interval (QTc) in range of 450 to less than 480 millisecond (msec), Maximum QTcB interval (Bazett's Correction) (msec) in range of 450 to less than 480 msec, Maximum QTcF interval (Fridericia's Correction) in range of 450 to less than 480 msec, maximum QTc interval increase from baseline in range of 30 to less than 60 msec and >=60 msec.
Time Frame: Baseline up to Week 16
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 30 | 33 | 32
Participants | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) Response
Description: Human serum ADA samples were analyzed for the presence or absence of anti--tanezumab antibodies by using a semi quantitative enzyme -linked immunosorbent assay (ELISA). Participants tested positive for ADA response on at least one post-baseline visit were reported. Participants with ADA titer level >=4.32 for PF-04383119 were considered as ADA positive.
Time Frame: Baseline up to Week 16
Population: Safety analysis population included all participants who received the day 1 IV infusion (either tanezumab or placebo infusion). Safety analysis population included all participants who received the day 1 IV infusion (either tanezumab or placebo infusion). Data for this outcome measure was not planned to be assessed collected and reported only for Tanezumab 50, 200 mcg/kg reporting group, not for placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

28. Secondary Outcome: Change From Baseline in Hopkins Verbal Learning Test - Revised (HVLT-R) at Week 2, 6, 12, 16 and End of Study
Description: HVLT-R was a word-list learning and memory test used to assess the changes in memory. The task was repeated, for a total of 3 learning trials. After a delay interval of 20 to 25 minutes, delayed recall trial was administered. 1)Learning efficiency: Assessed by examining the learning curve over 3 learning trials and by evaluating the sum of the scores for all 3 learning trials. Raw scores for each of the 3 learning trials were summed for the total recall (TR) score. The TR score ranges from 0 to 36, where higher scores indicated greater verbal learning and recall, 2) Ability to access newly learned information: Assessed by the number of words retained on the delayed recall (DR) trial and the percentage of words recalled from the word list. DR trial score ranges from 0 to 12, where higher scores indicated greater verbal learning and recall.
Time Frame: Baseline, Week 2, 6, 12, 16, end of study (i.e. anytime up to Week 16)
Population: Safety analysis population included all participants who received the day 1 IV infusion (either tanezumab or placebo infusion). Here, "number analyzed" signifies those participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Baseline: TR | 24.58 (3.59) | 23.15 (5.28) | 26.84 (5.54)
  Change at Week 2: TR: number analyzed (Participants) | 31 | 32 | 30
  Change at Week 2: TR | -0.03 (4.31) | 0.19 (3.73) | 0.70 (4.20)
  Change at Week 6: TR: number analyzed (Participants) | 22 | 29 | 26
  Change at Week 6: TR | 1.50 (5.02) | 0.83 (4.29) | 1.08 (3.86)
  Change at Week 12: TR: number analyzed (Participants) | 22 | 26 | 25
  Change at Week 12: TR | 2.18 (3.92) | 1.35 (4.43) | 1.56 (3.85)
  Change at Week 16: TR: number analyzed (Participants) | 21 | 27 | 23
  Change at Week 16: TR | 3.10 (4.35) | 1.93 (4.58) | 2.61 (3.43)
  End of Study: TR: number analyzed (Participants) | 31 | 32 | 30
  End of Study: TR | 3.03 (4.35) | 1.19 (4.71) | 2.37 (3.68)
  Baseline: DR | 9.16 (2.34) | 7.70 (2.48) | 9.47 (2.55)
  Change at Week 2: DR: number analyzed (Participants) | 30 | 32 | 30
  Change at Week 2: DR | -0.20 (2.34) | 0.63 (1.96) | 0.67 (1.42)
  Change at Week 6: DR: number analyzed (Participants) | 22 | 28 | 26
  Change at Week 6: DR | 0.09 (1.97) | 0.86 (2.10) | 0.85 (1.62)
  Change at Week 12: DR: number analyzed (Participants) | 22 | 26 | 25
  Change at Week 12: DR | 0.50 (1.95) | 1.23 (2.29) | 0.56 (1.87)
  Change at Week 16: DR: number analyzed (Participants) | 21 | 27 | 25
  Change at Week 16: DR | 1.10 (2.43) | 1.81 (3.08) | 1.09 (1.98)
  Change at End of study: DR: number analyzed (Participants) | 31 | 32 | 30
  Change at End of study: DR | 0.71 (2.55) | 1.69 (3.05) | 0.77 (1.92)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 2 (Learning): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.548, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.12, 90% CI 2-sided [-1.81 to 1.56], Standard Error of Mean 1.02
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.117, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 1.24, 90% CI 2-sided [-0.48 to 2.96], Standard Error of Mean 1.04
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 6 (Learning): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.779, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.86, 90% CI 2-sided [-2.69 to 0.98], Standard Error of Mean 1.11
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 28, analysis 3]; Test type: Superiority; p = 0.375, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.36, 90% CI 2-sided [-1.52 to 2.25], Standard Error of Mean 1.14
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 12 (Learning): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.881, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -1.36, 90% CI 2-sided [-3.26 to 0.54], Standard Error of Mean 1.15
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 28, analysis 5]; Test type: Superiority; p = 0.636, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -0.41, 90% CI 2-sided [-2.33 to 1.52], Standard Error of Mean 1.17
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 16 (Learning): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.905, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = -1.54, 90% CI 2-sided [-3.46 to 0.39], Standard Error of Mean 1.17
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 28, analysis 7]; Test type: Superiority; p = 0.499, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.00, 90% CI 2-sided [-2.00 to 2.00], Standard Error of Mean 1.21
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 2 (Delayed): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.297, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.27, 90% CI 2-sided [-0.56 to 1.09], Standard Error of Mean 0.50
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 28, analysis 9]; Test type: Superiority; p = 0.035, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.91, 90% CI 2-sided [0.09 to 1.74], Standard Error of Mean 0.50
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 6 (Delayed): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.222, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.41, 90% CI 2-sided [-0.48 to 1.31], Standard Error of Mean 0.54
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 28, analysis 11]; Test type: Superiority; p = 0.069, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.81, 90% CI 2-sided [-0.09 to 1.70], Standard Error of Mean 0.54
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 12 (Delayed): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.338, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.23, 90% CI 2-sided [-0.68 to 1.15], Standard Error of Mean 0.55
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 28, analysis 13]; Test type: Superiority; p = 0.381, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.17, 90% CI 2-sided [-0.75 to 1.09], Standard Error of Mean 0.56
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 50 mcg/kg; Week 16 (Delayed): LS Mean Difference was estimated from the repeated measures model with participant as random effect; treatment, week and treatment-by-week interaction as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.306, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.29, 90% CI 2-sided [-0.64 to 1.21], Standard Error of Mean 0.56
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 200 mcg/kg; [analysis description as in outcome 28, analysis 15]; Test type: Superiority; p = 0.440, Repeated Measures Model; P-value was based on repeated measures model from pairwise comparisons, and was 1-sided; LS Mean Difference = 0.09, 90% CI 2-sided [-0.87 to 1.04], Standard Error of Mean 0.58

29. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) for Tanezumab
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: Predose (0 hour) and 1, 2, 192, 193, 672, 673, 1008, 1009, 2016, 2017 and 2688 hours post dose on Day 1
Population: Pharmacokinetic (PK) analysis population included all participants who had at least 1 dose of study medication. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for placebo group.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 26 | 26
nanogram*hour per milliliter (ng*hr/mL) | 843814.9 (514324.95) | 2559793.7 (1332736.95)

30. Other Pre Specified Outcome: Area Under the Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) for Tanezumab
Description: Area under the plasma concentration time-curve from time zero to the time of last measured concentration (AUClast).
Time Frame: Predose (0 hour) and 1, 2, 192, 193, 672, 673, 1008, 1009, 2016, 2017 and 2688 hours post dose on Day 1
Population: PK analysis population included all participants who had at least 1 dose of study medication. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for placebo group.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 32 | 30
ng*hr/mL | 873666.5 (963283.79) | 2242378.0 (1128330.22)

31. Other Pre Specified Outcome: Plasma Concentration of Tanezumab at Nominal Collection Time of 1 Hours and 2688 Hours Postdose
Description: Plasma concentration of tanezumab at nominal collection time of 1 hour post-dose (C1) and plasma concentration at nominal collection time of 2688 hours post-dose (C2688) were reported.
Time Frame: 1, 2688 hours postdose on Day 1
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 33 | 32
nanogram per milliliter
  C1: number analyzed (Participants) | 32 | 30
  C1 | 2101.8 (1765.97) | 6861.6 (4885.51)
  C2688: number analyzed (Participants) | 31 | 25
  C2688 | 101.810 (325.241) | 170.984 (241.639)

32. Other Pre Specified Outcome: Total Clearance of Tanezumab From Plasma
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. It was calculated by dividing given intravenous dose by AUC inf. AUC inf is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: Predose (0 hour) and 1, 2, 192, 193, 672, 673, 1008, 1009, 2016, 2017 and 2688 hours post dose on Day 1
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: milliliter per hour per kilogram
Arm/Group | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 26 | 26
milliliter per hour per kilogram | 0.082 (0.053) | 0.093 (0.042)

33. Other Pre Specified Outcome: Terminal Elimination Half-Life (t1/2) of Tanezumab
Description: Terminal elimination half-life is the time measured for the plasma concentration of tanezumab to decrease by one half of its original concentration.
Time Frame: Predose (0 hour) and 1, 2, 192, 193, 672, 673, 1008, 1009, 2016, 2017 and 2688 hours post dose on Day 1
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 26 | 26
days | 18.92 (4.889) | 22.76 (7.336)

34. Other Pre Specified Outcome: Volume of Distribution at Steady State (Vss) for Tanezumab
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: Predose (0 hour) and 1, 2, 192, 193, 672, 673, 1008, 1009, 2016, 2017 and 2688 hours post dose on Day 1
Population: PK analysis population included all participants who had at least 1 dose of study medication. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed placebo group.
Measure: Mean (Standard Deviation); unit: milliliter per kilogram
Arm/Group | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 26 | 26
milliliter per kilogram | 47.03 (22.334) | 65.96 (18.785)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | Tanezumab 50 mcg/kg | Tanezumab 200 mcg/kg
Serious Adverse Events (participants affected / at risk) | 1/31 | 2/33 | 1/32
Other Adverse Events (participants affected / at risk) | 20/31 | 24/33 | 21/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Tanezumab 50 mcg/kg (N=33) | Tanezumab 200 mcg/kg (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Tanezumab 50 mcg/kg (N=33) | Tanezumab 200 mcg/kg (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 2 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 1
Mastitis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 3
Viral infection (Infections and infestations) | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase abnormal (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 2 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 4
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Intention tremor (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 3
Presyncope (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.